CLINICAL TRIAL: NCT02815904
Title: Effects of Early Yakson Touch and Kinesthetic Stimulation on the Development of High Risk neonates-a Randomized Controlled Trial
Brief Title: Effects of Early Yakson Touch and Kinesthetic Stimulation on the Development of High Risk Neonates
Acronym: YTKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Assistant Professor, Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMU/IEC/2016/751; U1111-1184-4324 (Other: Universal Trial Number (UTN)); 2016-002659-29 (EudraCT Number)
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Preterm Infants; Infant, Low Birth Weight
Keywords: Neonates; physical therapy; neonatal intensive care units; yakson touch; kinesthetic stimulation
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yakson touch and Kinesthetic stimulation (Experimental): Yakson touch (YT) The therapist will relax arms and shoulder muscles for 1 minute and will do deep breathing to accumulate Ki energy on the palms. The Therapist will apply Yakson on the neonate.
  Kinesthetic stimulation (KS) For giving kinesthetic stimulation the neonate will be placed in supine position. There will be six passive flexion and extension movements. Each of the movement will each last for approximately 10 seconds. The movements will be performed in the following order -right arm, left arm, right leg, left leg, both legs simultaneously
  Interventions: Other: Yakson touch; Other: Kinesthetic stimulation
- Conventional Handling and KMC (Active Comparator): Conventional Handling (CH) The neonates in control group will receive developmental positioning(positioning of preterm infants for optimal physiological development) for 20 minutes per hour for 5 days.
  Kangaroo mother care (KMC) Holding the neonate skin to skin by mother for one hour a day
  Interventions: Other: Conventional handling; Other: Kangaroo Mother Care

INTERVENTIONS:
Other: Yakson touch — Yakson is a Korean therapeutic touch given to neonates and infants by caressing their abdomen with one hand while the other hand is placed on the back of the neonate\infant to relieve their pain or to calm them down.
  Other Names: YT
  Arms: Yakson touch and Kinesthetic stimulation
Other: Conventional handling — Positioning of preterm infants for optimal physiological development
  Other Names: CH
  Arms: Conventional Handling and KMC
Other: Kinesthetic stimulation — For kinesthetic stimulation, all the limbs were given six passive flexion and extension movements
  Other Names: KS
  Arms: Yakson touch and Kinesthetic stimulation
Other: Kangaroo Mother Care — Providing skin to skin human touch
  Other Names: KMC
  Arms: Conventional Handling and KMC

SUMMARY:
The role of physiotherapy interventions in treatment of high risk infants has not been established even after a number of studies. The high risk infants are prone to developmental delays and early intervention is most effective for them owing to the plasticity of brain in early infancy. Yakson is one among the most effective and safe methods of tactile stimulation for preterm neonates. Tactile and kinesthetic stimulation techniques have been proved to be effective but there is no standardized protocol. The present study will try to investigate the efficacy of Yakson touch in combination with kinesthetic stimulation on the development of high risk neonates against conventional handling which will include developmental positioning and Kangaroo mother care.

DETAILED DESCRIPTION:
Yakson touch

1. Universal precautions to maintain sterile conditions will be taken.
2. Then the therapist will warm both hands with a radiant warmer so that the temperature of the palms reaches between 93F and 94F (33.9-34.4°C). Digital thermometer will be used to check the temperature of palms.
3. The therapist will relax arms and shoulder muscles for 1 minute and will do deep breathing to accumulate Ki energy on the palms.
4. The Therapist will apply Yakson on the neonate. Yakson will be given for 15 minutes which will be divided into resting the hands, caressing gently, and again resting the hands, each of which will last for 5 minutes. Throughout the application of Yakson, fingers and palm of the therapist will be in constant contact and the contact will be such that there is no pressure on the infant.
5. Resting the hands for 5 minutes- While one hand is resting on the chest and abdomen of the neonate and other hand is supporting the back, the therapist will concentrate on resting hands assuming that a healthy Ki energy is passing to the neonate. During this therapist will do slow breathing to remain relaxed.
6. Caressing gently for 5 minutes-With hand in same position, the therapist will caress repeatedly for 5 minutes. Therapist will caress for 1 minute, rest for 30 seconds, caress for 1 minute, rest for 30 seconds and caress for 2 minutes. The therapist will caress the abdomen and chest of the infant in clockwise direction in a diameter of 1 centimeter in circular motion every 10 seconds
7. Resting the hands for 5 minutes- The therapist will rest the hands as previously described.

(* The therapist will caress repeatedly for 5 minutes. Therapist will caress for 1 minute, rest for 30 seconds, caress for 1 minute, rest for 30 seconds and caress for 2 minutes. The therapist will caress the abdomen and chest of the infant in clockwise direction in a diameter of 1 centimeter in circular motion every 10 seconds.)

Kinesthetic stimulation For giving kinesthetic stimulation the infant will be placed in supine position. There will be six passive flexion and extension movements. Each of the movement will each last for approximately 10 seconds. The movements will be performed in the following order -right arm, left arm, right leg, left leg, both legs simultaneously

Control group treatment The neonates in control group will receive Kangaroo mother care (holding the neonate skin to skin by mother) for one hour a day and developmental positioning(positioning of preterm infants for optimal physiological development) for 20 minutes per hour for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with birth weight less than 2500 grams and born before 37 weeks of gestation males and females will be recruited in the study

Exclusion Criteria:

* Medically unstable neonates or neonates with communicable disease or congenital anomaly or skin infection will be excluded from the study

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Neonatal behavioral assessment scale (NBAS) | Change from Baseline Neonatal behavioral assessment scale at 1 week
  Neonatal behavioral assessment scale (NBAS) will be used to monitor the effects of Yakson touch and kinesthetic stimulation on the development of high risk neonates. Baseline reading of NBAS will be recorded for the neonates in control and experimental groups before the beginning of intervention. The NBAS contains 28 behavioural items, 18 reflex items, and 7 supplementary items for fragile or high-risk infants. It is a neurobehavioural screening tool

SECONDARY OUTCOMES:
Heart rate | up to 1 week
  Recorded pre and post intervention for each session
Respiratory rate | up to 1 week
  Recorded pre and post intervention for each session
Systolic Blood Pressure | up to 1 week
  Recorded pre and post intervention for each session
Saturation of inhaled oxygen | up to 1 week
  Recorded pre and post intervention for each session

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Parashar, BPT, Principal Investigator — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, Maharishi Markandeshwar University
Locations (1):
- Preeti Parashar, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Parashar P, Samuel AJ, Aranha VP. Efficacy of early Yakson touch and kinaesthetic stimulation (YAKIN) on the development of high risk neonates: A randomized controlled trial protocol. J Nepal Paediatr Soc 2017;37(2):173-9.
Supporting Information: Study Protocol
Time Frame: Published in, Journal of Nepal Paediatric Society
Access Criteria: Full-text available free at the journal site
URL: http://dx.doi.org/10.3126/jnps.v37i2.16724

REFERENCES:
- [Background] Bahman Bijari B, Iranmanesh S, Eshghi F, Baneshi MR. Gentle Human Touch and Yakson: The Effect on Preterm's Behavioral Reactions. ISRN Nurs. 2012;2012:750363. doi: 10.5402/2012/750363. Epub 2012 Jun 25. PMID 22792482
- [Background] Pillai Riddell RR, Racine NM, Turcotte K, Uman LS, Horton RE, Din Osmun L, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Gerwitz-Stern A. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD006275. doi: 10.1002/14651858.CD006275.pub2. PMID 21975752
- [Background] Im H, Kim E, Park E, Sung K, Oh W. Pain reduction of heel stick in neonates: Yakson compared to non-nutritive sucking. J Trop Pediatr. 2008 Feb;54(1):31-5. doi: 10.1093/tropej/fmm083. Epub 2007 Oct 25. PMID 17962243
- [Background] Im H, Kim E. Effect of Yakson and Gentle Human Touch versus usual care on urine stress hormones and behaviors in preterm infants: a quasi-experimental study. Int J Nurs Stud. 2009 Apr;46(4):450-8. doi: 10.1016/j.ijnurstu.2008.01.009. Epub 2008 Mar 18. PMID 18353332
- [Background] Im H, Kim E, Cain KC. Acute effects of Yakson and Gentle Human Touch on the behavioral state of preterm infants. J Child Health Care. 2009 Sep;13(3):212-26. doi: 10.1177/1367493509337441. PMID 19713405